CLINICAL TRIAL: NCT06590688
Title: Extracellular Water for Volume Status Characterization in Patients with Intracranial Hemorrhage
Brief Title: Defining Volume Status with Extracellular Water Measurement in Patients with Intracranial Hemorrhage
Status: Not yet recruiting | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-06866-01.3
Record Dates: First submitted 2024-07-18; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Intracranial Hemorrhages
MeSH Terms: conditions — Intracranial Hemorrhages

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples With DNA — Blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to learn about the influence of extracellular water on volume status in adult patients with intracranial hemorrhage presenting with hemodynamic instability. The main question it aims to answer is:

• Can measurement of extracellular water contribute to the description of hemodynamic instability in adult patients with intracranial hemorrhage. Patients with intracranial hemorrhage admitted to intensive care will receive standard care with the addition of measurement of extracellular water.

DETAILED DESCRIPTION:
Adult patients with intracranial hemorrhage admitted to ICU will be recruited. During the first five days after inclusion blood samples and extended non-invasive monitoring, including monitoring of the microcirculation (CytoCam) and measurement of extracellular water (dielectronic constant), will be added to routine care and monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Adults with intracranial hemorrhage admitted to ICU.

Exclusion Criteria:

* Pregnancy, palliative care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to ICU in Uppsala with intracranial hemorrhage.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-09-23 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Extracellular water for volume status characterization in patients with intracranial hemorrhage. | 7 days
  Can measurement of extracellular water (MoistureMeterD, Delfin Technologies Ltd, Kuopio, Finland) contribute to the description of hemodynamic instability in adult patients with intracranial hemorrhage during the first five days?

CONTACTS AND LOCATIONS:
Overall Officials: Annelie Barrueta Tenhunen, Principal Investigator — Uppsala University, Region Uppsala

IPD SHARING:
Plan to Share IPD: No
The data will only be accessible to the research team.

REFERENCES:
- [Background] Nuutinen J, Ikaheimo R, Lahtinen T. Validation of a new dielectric device to assess changes of tissue water in skin and subcutaneous fat. Physiol Meas. 2004 Apr;25(2):447-54. doi: 10.1088/0967-3334/25/2/004. PMID 15132310
- [Background] Toro C, Markarian B, Mayrovitz HN. Breast Cancer-Related Lymphedema Assessed via Tissue Dielectric Constant Measurements. Cureus. 2024 Apr 29;16(4):e59261. doi: 10.7759/cureus.59261. eCollection 2024 Apr. PMID 38813316
- [Background] Gress DR; Participants in the International Multi-Disciplinary Consensus Conference on the Critical Care Management of Subarachnoid Hemorrhage. Monitoring of volume status after subarachnoid hemorrhage. Neurocrit Care. 2011 Sep;15(2):270-4. doi: 10.1007/s12028-011-9604-x. PMID 21751101